CLINICAL TRIAL: NCT01613755
Title: The Effect of Dipyridamole on the Pharmacokinetics of Metformin
Brief Title: Metformin-Dipyridamole Interaction Trial
Acronym: MetDipy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Met-Dipy001
Record Dates: First submitted 2012-05-25; First posted 2012-06-07 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes
Keywords: Effect Dipyridamole on pharmacokinetics of metformin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin; Dipyridamole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin therapy with concomitant use of dipyridamole (Active Comparator): Metformin 500 mg twice daily for four days in combination with dipyridamole 200 mg twice daily for four days
  Interventions: Drug: Metformin, dipyridamole
- Metformin therapy (Active Comparator): Metformin 500 mg twice daily for four days
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin, dipyridamole — Metformin 500 mg twice daily for four days Dipyridamole 200 mg twice daily for four days
  Arms: Metformin therapy with concomitant use of dipyridamole
Drug: Metformin — Metformin 500 mg twice daily for four days
  Arms: Metformin therapy

SUMMARY:
The antihyperglycemic drug metformin and the thrombocyte aggregation inhibitor dipyridamole are often used concomitantly in patients with diabetes who have suffered a transient ischemic attack or stroke. It has recently been suggested that the gastrointestinal absorption of metformin is mediated by the equilibrative nucleoside transporter 4 (hENT4). Dipyridamole has been reported to inhibit hENT4 transport in vitro. The aim of this research proposal is to study the pharmacokinetic interaction between metformin and dipyridamole. The investigators hypothesize that dipyridamole reduces the gastrointestinal absorption of metformin. If this hypothesis can be confirmed, then the results of this study can explain in part the high variability in plasma metformin concentrations in patients treated with diabetes, and can be used to optimize pharmacotherapy in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Written informed consent

Exclusion Criteria:

* Smoking
* Hypertension (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg)
* Diabetes Mellitus (fasting glucose >7.0 mmol/L or random glucose >11 mmol/L)
* History of any cardiovascular disease
* Concomitant use of medication
* Renal dysfunction (MDRD <60 ml/min)
* ECG abnormalities, other than firs grade AV-block or right bundle branch block

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The area under the curve of the metformin plasma concentration at several timepoints | 10 hours after ingestion of last dose of metformin
  The area under the curve of the metformin plasma concentration at t=0, t=1, t=2, t=2.5, t=3, t=3.5, t=4, t=5, t=6, t=8, and t=10 hours after the intake and the Cmax.
Peak plasma concentration (Cmax) of metformin | about 3 hours after intake of last dose of metformin
  Peak plasma concentration (Cmax) of metformin

CONTACTS AND LOCATIONS:
Overall Officials: N. Riksen, MD, PhD, Principal Investigator — Radboud University Medical Center; G. Rongen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands